CLINICAL TRIAL: NCT06269848
Title: Talent Identification in Young Boxers Form the State of Mexico
Brief Title: Identification of Sports Talents in Boxers
Status: Active, not recruiting | Type: Observational
Sponsor: Dynamical Business and Science Society - DBSS International SAS (Network)
Responsible Party: Sponsor
Other Study IDs: ITaDeBo
Record Dates: First submitted 2024-01-19; First posted 2024-02-21 (Actual); Last update posted 2024-03-01 (Actual); Status verified 2024-02

CONDITIONS: Body Composition; Exercise Test; Psychological Well-Being
Keywords: Boxing; Talent selection; Youths; Sport; Mexicans
MeSH Terms: conditions — Psychological Well-Being

STUDY DESIGN:
Observational Model: Other | Time Perspective: Cross-Sectional
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (2):
- Junior boxers: Junior category boxers aged 15 to 16 years old
- Youth boxers: Youth category boxers aged 17 to 18 years old

SUMMARY:
This study aims to identify sporting talents by profiling a group of young boxers residing in the State of Mexico using unsupervised machine learning methods. This study is supported by Asociación de Boxeo del Estado de México AC (ABEM) and powered by DBSS.

DETAILED DESCRIPTION:
This cross-sectional study aims to identify sporting talents by profiling a group of young boxers residing in the State of Mexico. The primary outcomes encompass anthropometric, physical, and psychological variables associated with sports performance. In detail, a morphological and body composition analysis will be conducted using anthropometric data. Boxing performance will be assessed by measuring the average acceleration of straight punches over 6 seconds, impact force in the straight boxing punch using a load cell, reactive force index in a counter-movement jump on a force platform, maximum isometric strength in the mid-thigh isometric pull on a force platform, load-velocity profile in the squat exercise using a linear encoder, and cardiorespiratory fitness measured with digital spirometry. Psychometric variables will include well-being level calculated with PERMA+4, attention capacity, perceptual acuity, concentration using the Toulouse test, and coping mechanisms assessed through the coping modes scale.

ELIGIBILITY:
Inclusion Criteria: Amateur boxers from the State of Mexico with no declared health issues -

Exclusion Criteria: Amateur boxers from the State of Mexico with any declared health issues

-

Ages: 15 Years to 18 Years | Sex: All
Age Groups: Child, Adult
Study Population: Amateur boxers from the State of Mexico, aged between 15 to 18 years, who will participate in the qualifying tournament for the 2024 national boxing championship organized by the Mexican Boxing Federation.
Sampling Method: Non-Probability Sample
Enrollment: 178 (Actual)
Dates: Start 2024-02-29 (Actual); Primary Completion 2024-03-11 (Estimated); Study Completion 2024-06-30 (Estimated)

PRIMARY OUTCOMES:
Anthropometry-Based Analysis of Adiposity | 10-15 minutes
  Anthropometric measurements will be carried out to estimate body composition, following the protocol established by the International Society for the Advancement of Kinanthropometry (ISAK). The absolute values of the sum of skinfolds (∑S) and related variables, such as skinfold-corrected girths, will be used for measuring adiposity.
The acceleration of the fists in straight boxing punches | <1 minutes
  Corner brand accelerometers will be used to measure the acceleration of the fists during the execution of repeated straight punches over a period of 6 seconds
Number of punches thrown within a specific timeframe | <1 minutes
  Corner brand accelerometers will be used to measure the quantity of straight punches performed within a 6-second timeframe.
Punch impact force | <1 minutes
  A load cell placed within a damping device will be used to measure the force applied after a straight boxing punch.
Reactive force index | <2 minutes
  A force platform will be used to measure the lower-limbs reactive force index during a countermovement jump (CMJ)
Cardiorespiratory fitness | <3 minutes
  A digital spirometry will be performed to measure the lung capacity of the participants. The Forced Expiratory Volume in the first second (FEV1) and Forced Vital Capacity (FVC) will be registered. Subsequently, the ratio FEV1/FVC will be calculated to obtain the percentage of forced vital capacity expelled in the first second.
Isometric Mid-Thigh Pull | <1 minutes
  The participants' force production capacity will be assessed. The test will be conducted on a force platform.
Load-velocity profile | <5 minutes
  To estimate the load-velocity profile, the two-point method can be used, where two loads corresponding approximately to 40-50% and 70-80% of the one-repetition maximum (RM) for the squat exercise are employed. The velocity of the load is measured in each attempt. This approach provides a reliable alternative for evaluating muscle mechanical capabilities through the relationship of the load-velocity profile, which aids in predicting Maximum Dynamic Strength. Moreover, it can be a quick and secure method for predicting this parameter in various exercises.

SECONDARY OUTCOMES:
Well-being profile | 5 minutes
  The PERMA+4 questionnaire will be administered to assess the well-being of the participants. The 10 circles in each domain represent a scale for evaluating well-being, where 1 is Completely Disagree and 10 is Completely Agree. A combined score is computed to report results.
Ways of Coping Questionnaire | <1 hour
  The coping modes scale consists of 66 items, which are statements regarding coping strategies, addressing both emotion and problem-solving. Response options range from 0 to 3, where 0 corresponds to 'Not at all' and 3 to 'To a great extent.' The scales will be administered to participants at the camp during a relaxation period away from physical tests.
Attention and Perceptual Processes | 10 minutes
  The Toulouse Test will be administered to measure individuals' attention capacity, perceptual acuity, concentration, as well as their resistance to monotony.

CONTACTS AND LOCATIONS:
Overall Officials: Ivan Ávila Castro, Lic., Study Chair — Círculo Internacional de Expertos en Deportes de Combate; Diego A Bonilla, Study Director — Research Division, Dynamical Business & Science Society-DBSS International SAS; Rodrigo D Merlo, PhD, Principal Investigator — Escuela Nacional de Entrenadores Deportivos; Juan A Rodríguez Chávez, Mg., Study Chair — Research Division, Dynamical Business & Science Society-DBSS International SAS; Jorge L Petro, Study Chair — Research Division, Dynamical Business & Science Society-DBSS International SAS; Augusto H Tardito, Lic., Study Chair — Círculo Internacional de Expertos en Deportes de Combate
Locations (1):
- Centro Ceremonial Otomí, México, Mexico

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Result] Finlay MJ, Page RM, Greig M, Bridge CA. Test-retest reliability and sensitivity of senior elite amateur boxers maximal punch force, as quantified by a vertically mounted force plate. PLoS One. 2023 Aug 10;18(8):e0289791. doi: 10.1371/journal.pone.0289791. eCollection 2023. PMID 37561692
- [Result] Loturco I, McGuigan MR, Pereira LA, Pareja-Blanco F. The load-velocity relationship in the jump squat exercise. Biol Sport. 2023 Apr;40(2):611-614. doi: 10.5114/biolsport.2023.118019. Epub 2022 Sep 6. PMID 37077791
- [Result] Merlo R, Rodriguez-Chavez A, Gomez-Castaneda PE, Rojas-Jaramillo A, Petro JL, Kreider RB, Bonilla DA. Profiling the Physical Performance of Young Boxers with Unsupervised Machine Learning: A Cross-Sectional Study. Sports (Basel). 2023 Jul 7;11(7):131. doi: 10.3390/sports11070131. PMID 37505618
- [Result] Bonilla DA, De Leon LG, Alexander-Cortez P, Odriozola-Martinez A, Herrera-Amante CA, Vargas-Molina S, Petro JL. Simple anthropometry-based calculations to monitor body composition in athletes: Scoping review and reference values. Nutr Health. 2022 Mar;28(1):95-109. doi: 10.1177/02601060211002941. Epub 2021 Apr 1. PMID 33792415